CLINICAL TRIAL: NCT00411892
Title: Effect of Inhaled Insulin (AERx® iDMS) Plus Pioglitazone Versus Pioglitazone Alone on HbA1c in Subjects With Type 2 Diabetes
Brief Title: Effect of Inhaled Insulin (AERx® iDMS) on Blood Glucose Control in Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-1683
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: pioglitazone; Drug: inhaled human insulin
- B (Active Comparator)
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: pioglitazone — Tablets, 45 mg/day.
Drug: inhaled human insulin — Treat-to-target dose titration scheme, inhalation.
  Other Names: NN1998
  Arms: A

SUMMARY:
This trial is conducted in the United States of America (USA). This trial will compare the changes in HbA1c after 26 weeks of inhaled insulin and pioglitazone combination therapy versus pioglitazone treatment alone.

DETAILED DESCRIPTION:
The decision to discontinue the development of AERx® is not due to any safety concerns. An analysis concluded that fast-acting inhaled insulin in the form it is known today, is unlikely to offer significant clinical or convenience benefits over injections of modern insulin with pen devices.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Current treatment with oral antidiabetes drugs (OADs) for at least 2 months
* HbA1c between 7.0-11.0% if on OAD monotherapy
* HbA1c between 7.0-10.0% if on OAD combination therapy
* BMI less than or equal to 40 kg/m2

Exclusion Criteria:

* Current regular smoking or regular smoking within the last 6 months
* Current acute or chronic pulmonary disease (except for asthma)
* Proliferative retinopathy requiring treatment
* Clinically significant disease history including kidney or liver disease, or heart disease which limits physical activity or results in discomfort with physical activity
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2006-11-29 (Actual); Primary Completion 2008-03-18 (Actual); Study Completion 2008-03-18 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline | After 26 weeks of treatment

SECONDARY OUTCOMES:
Fasting plasma glucose | after 26 weeks of treatment
Lipid profiles | after 26 weeks of treatment
Frequency of hypoglycaemic episodes | after 26 weeks of treatment
Glucose profiles | at pre- and post meals, bedtime and 3:00 am
Change in body weight | after 26 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (103):
- United States (103):
  - Novo Nordisk Investigational Site, Ozark, Alabama
  - Novo Nordisk Investigational Site, Tuscaloosa, Alabama
  - Novo Nordisk Investigational Site, Vestavia Hills, Alabama
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Bermuda Dunes, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Roseville, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Santa Barbara, California
  - Novo Nordisk Investigational Site, Temecula, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Arvada, Colorado
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Beverly Hills, Florida
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Marianna, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Niceville, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Panama City, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Vero Beach, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Blue Ridge, Georgia
  - Novo Nordisk Investigational Site, Dunwoody, Georgia
  - Novo Nordisk Investigational Site, Powder Springs, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Sandy Springs, Georgia
  - Novo Nordisk Investigational Site, Suwanee, Georgia
  - Novo Nordisk Investigational Site, Tucker, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Avon, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Lafayette, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Prince Frederick, Maryland
  - Novo Nordisk Investigational Site, Marlborough, Massachusetts
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Bloomington, Minnesota
  - Novo Nordisk Investigational Site, Jackson, Mississippi
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, High Point, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Bismarck, North Dakota
  - Novo Nordisk Investigational Site, Canal Fulton, Ohio
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Clinton, Oklahoma
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Bensalem, Pennsylvania
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Clarksville, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Lewisville, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Arlington, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Warrenton, Virginia
  - Novo Nordisk Investigational Site, Tacoma, Washington

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com